CLINICAL TRIAL: NCT05452291
Title: Exploring Multiomics Biomarkers for Urolithiasis
Brief Title: Multiomics Biomarkers for Urolithiasis
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2022.093
Record Dates: First submitted 2022-06-27; First posted 2022-07-11 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective case series study. To compare urine sample of recurrent stone-formers and non-stone former by multiomics approach to identify potential markers for stone recurrence.

DETAILED DESCRIPTION:
A total of 100 Chinese patients with history of recurrent urinary stone and no history of urinary stone disease (control) will be recruited for the study.

Urine will be saved for multiomics analysis, including metabolomics, proteomics, etc. Thereafter, integrated multiomics calculation of recurrent stone can be studied for the differentiation of recurrent stone former and non-stone former.

After completing the preliminary and screening experiments, a large validation cohort (1000 Chinese patients with history of recurrent urinary stone) will be carried out. The patients will then be follow-up in clinic for at least 3 years, with minimum annual review and imaging to detect for any stone recurrence, as defined as increase in stone size and number, or symptomatic stone events. Targeted biomarkers measurement, based on part 1 result, will be done and the result will be used to correlated with the clinical outcomes of stone recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of recurrent urinary stone
* Age greater than or equal to 18 years old
* Have more than 2 episodes of radio-opaque stone disease (bilateral stones were counted as two episode)

Patients with no history of urinary stone disease

* Age greater than or equal to 18 years old
* With no history of urinary calculi, from history and imaging.

Exclusion criteria:

* Patient refused or unable to provide consent for the study
* Patient with active urinary infection
* Patient with radiolucent stone or infective stone
* Patients with no history of urinary stone disease (for control group)
* Patient refused or unable to provide consent for the study
* Patient with active urinary infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects have more than 2 episodes of radio-opaque stone disease
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Level of urinary metabolomics by multiomics approach in non-stone former | every year up to 3 year
  Patient will be reviewed with urine collection for the level of urinary metabolomics including metabolomics and proteomics by multiomics analysis every year up to 3 years
Change of Level of urinary proteomics by multiomics approach in recurrent stone-formers | every year up to 3 year
  Patient will be reviewed with urine collection for the level of urinary metabolomics including metabolomics and proteomics by multiomics analysis and there will be radiological imaging annually to check if there is any suspect stone every year up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singal RK, Denstedt JD. Contemporary management of ureteral stones. Urol Clin North Am. 1997 Feb;24(1):59-70. doi: 10.1016/s0094-0143(05)70354-2. PMID 9048852
- [Background] Netto Junior N, Claro JF, Ferreira U, Lemos GC. Lumbar ureteric stones: which is the best treatment? Urology. 1991 Nov;38(5):443-6. doi: 10.1016/0090-4295(91)80234-x. PMID 1949455
- [Background] Wong MY, Li MK, Foo KT. Extracorporeal shockwave lithotripsy using Storz Modulith SL20--the Singapore General Hospital experience. Ann Acad Med Singap. 1993 Nov;22(6):905-7. PMID 8129354
- [Background] Carr LK, D'A Honey J, Jewett MA, Ibanez D, Ryan M, Bombardier C. New stone formation: a comparison of extracorporeal shock wave lithotripsy and percutaneous nephrolithotomy. J Urol. 1996 May;155(5):1565-7. doi: 10.1016/s0022-5347(01)66127-5. PMID 8627823
- [Background] Segura JW, Preminger GM, Assimos DG, Dretler SP, Kahn RI, Lingeman JE, Macaluso JN Jr. Ureteral Stones Clinical Guidelines Panel summary report on the management of ureteral calculi. The American Urological Association. J Urol. 1997 Nov;158(5):1915-21. doi: 10.1016/s0022-5347(01)64173-9. PMID 9334635
- [Background] Yamada K, Tanokura M, Kawano Y. High-energy phosphate turnover in muscle contraction: time-resolved 31P NMR studies. Prog Clin Biol Res. 1989;315:185-95. No abstract available. PMID 2508132
- [Background] Kamihira O, Ono Y, Katoh N, Yamada S, Mizutani K, Ohshima S. Long-term stone recurrence rate after extracorporeal shock wave lithotripsy. J Urol. 1996 Oct;156(4):1267-71. PMID 8808851
- [Background] Eisner BH, Goldfarb DS. A nomogram for the prediction of kidney stone recurrence. J Am Soc Nephrol. 2014 Dec;25(12):2685-7. doi: 10.1681/ASN.2014060631. Epub 2014 Aug 7. No abstract available. PMID 25104802
- [Background] Schmid M, Dalela D, Tahbaz R, Langetepe J, Randazzo M, Dahlem R, Fisch M, Trinh QD, Chun FK. Novel biomarkers of acute kidney injury: Evaluation and evidence in urologic surgery. World J Nephrol. 2015 May 6;4(2):160-8. doi: 10.5527/wjn.v4.i2.160. PMID 25949930
- [Background] Alexandroff AB, Jackson AM, Chisholm GD, James K. Cytokine modulation of epidermal growth factor receptor expression on bladder cancer cells is not a major contributor to the antitumour activity of cytokines. Eur J Cancer. 1995 Nov;31A(12):2059-66. doi: 10.1016/0959-8049(95)00210-3. PMID 8562166
- [Background] Balbay D, Ozen H, Ozkardes H, Barut A, Bakkaloglu M, Tasar C, Remzi D. Detection of urinary interleukin-2, interleukin-2 receptor, and tumor necrosis factor levels in patients with superficial bladder tumors after intravesical BCG immunotherapy. Urology. 1994 Feb;43(2):187-90. doi: 10.1016/0090-4295(94)90042-6. PMID 8116114
- [Background] Shum DK, Gohel MD, Tam PC. Hyaluronans: crystallization-promoting activity and HPLC analysis of urinary excretion. J Am Soc Nephrol. 1999 Nov;10 Suppl 14:S397-403. PMID 10541272